CLINICAL TRIAL: NCT06787222
Title: Effectiveness and Safety of Zingiber Officinale Transdermal Patch for Acne Vulgaris; Study of Interleukin 1 and Skin Microbiome
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hasanuddin University (Other)
Responsible Party: Principal Investigator, Rini Amanda Carolina Saragih, Principle investigator, Hasanuddin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 700/UN4.6.4.5.31/PP36/2024
Record Dates: First submitted 2025-01-16; First posted 2025-01-22 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2024-11

CONDITIONS: Acne Vulgaris
Keywords: acne vulgaris, zingiber officinale, microbiome
MeSH Terms: conditions — Acne Vulgaris | interventions — Tretinoin

STUDY DESIGN:
Intervention Model Description: Researcher will compare both half faces (split face); one side as treatment side where patch is used, and another side as control. Patient will be asked to apply tretinoin 0,025% cream nightly. After applying tretinoin 0,025% on whole face, patient will be asked to apply patch on a pustule on one half face, and no patch will be used on another half face.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- tretinoin 0.025% + Z.officinale patch (Experimental): Z. officinale 0.05% application on pustule after tretinoin 0.025% application
  Interventions: Drug: tretinoin 0.025% + Z. officinale patch
- tretinoin 0.025% cream (Active Comparator): No Z. officinale patch
  Interventions: Drug: tretinoin 0.025% cream

INTERVENTIONS:
Drug: tretinoin 0.025% + Z. officinale patch — Material used for patch formulation were 3,15 grams of polyvinyl alcohol, 4,2 grams of polyvinyl pyrrolidone, 12,6 ml distilled water, and 1,05 grams of Z. officinale extract.
  Arms: tretinoin 0.025% + Z.officinale patch
Drug: tretinoin 0.025% cream — no Z. officinale patch applied after tretinoin 0.025% application
  Arms: tretinoin 0.025% cream

SUMMARY:
The goal of this clinical trial is to investigate the effectivity and safety of mild to moderate acne vulgaris therapy using Zingiber officinale 5 % transdermal patch. Researcher will compare both half faces (split face); one side as treatment side where patch is used, and another side as control. Patient will be asked to apply tretinoin 0,025% cream nightly. After applying tretinoin 0,025% on whole face, patient will be asked to apply patch on a pustule on one half face, and no patch will be used on another half face.

Total lesion count will be assessed before treatment and 21 days after treatment. Specimen for skin microbiome and interleukin examination will be collected before and 21 days after treatment.

DETAILED DESCRIPTION:
Current acne vulgaris treatment include antibiotic, retinoic acid, and benzoyl peroxide. The use of antibiotic has been linked to antibiotic resistant problem. Research also has shown the association between acne vulgaris and skin microbiome. Therefore, new treatment for acne vulgaris that has good effect on skin microbiome is needed.

Z. officinale is an herb that commonly used in traditional medicine. Researches have shown that it has anti-inflammation activity and antibiotic activity to Cutibacterium acnes. On the other hand, the prebiotic potency of Z. officinale on gut microbiome has also been investigated.

This randomized controlled trial shall include 26 mild to moderate acne vulgaris patients according to inclusion and exclusion criteria. Patches will be given every 5 days as researcher follow up patient condition. Patient photograph will be taken before treatment, on follow up day, and after 21 days treatment. Skin microbiome specimen will be collected using skin swab method. Secret from a chosen pustule will be collected for interleukin examination.

During clinical trial, patient will use non comedogenic sunscreen and soap from researcher. Patient will be asked to report to researcher if there is side effect of treatment.

ELIGIBILITY:
Inclusion Criteria:

* female
* 15-45 years old
* mild to moderate acne vulgaris according to Lehmann criteria
* minimal 3 pustules on face that are distributed on right and left sides

Exclusion Criteria:

* history of allergy to ingredients that is used in research
* history of topical acne medication and steroid in the last 2 weeks
* history of medical aesthetic procedure such as laser and chemical peeling in the last 2 weeks
* history of oral antibiotic therapy in the last 6 weeks
* history of oral isotretinoin therapy in the last 6 months
* history of probiotic consumption in the last 3 weeks
* pregnancy and lactation

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-11-03 (Actual); Primary Completion 2025-08-25 (Actual); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Total inflammatory acne lesions | At 0 and after 3 weeks duration of trial
  Total inflammatory acne lesions are the total of papules, pustules, nodules, and cysts.

SECONDARY OUTCOMES:
Level of Interleukin-1 from pustule | At 0 and after 3 weeks duration of trial
  Level of interleukin-1 will be measured using ELISA method
Skin microbiome | At 0 and after 3 weeks duration of trial
  S. epidermidis/ C. acnes ratio will be measured using digital Polymerase Chain Reaction

CONTACTS AND LOCATIONS:
Locations (1):
- Doctoral Programme, Faculty of Medicine, Hasanuddin University, Makassar, South Sulawesi, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang X, Zhang D, Jiang H, Zhang S, Pang X, Gao S, Zhang H, Zhang S, Xiao Q, Chen L, Wang S, Qi D, Li Y. Gut Microbiota Variation With Short-Term Intake of Ginger Juice on Human Health. Front Microbiol. 2021 Feb 23;11:576061. doi: 10.3389/fmicb.2020.576061. eCollection 2020. PMID 33708178
- [Background] Lebeer S, Oerlemans EFM, Claes I, Henkens T, Delanghe L, Wuyts S, Spacova I, van den Broek MFL, Tuyaerts I, Wittouck S, De Boeck I, Allonsius CN, Kiekens F, Lambert J. Selective targeting of skin pathobionts and inflammation with topically applied lactobacilli. Cell Rep Med. 2022 Feb 15;3(2):100521. doi: 10.1016/j.xcrm.2022.100521. eCollection 2022 Feb 15. PMID 35243421
- [Background] Wang X, Howe S, Deng F, Zhao J. Current Applications of Absolute Bacterial Quantification in Microbiome Studies and Decision-Making Regarding Different Biological Questions. Microorganisms. 2021 Aug 24;9(9):1797. doi: 10.3390/microorganisms9091797. PMID 34576694
- [Background] Byrd AL, Belkaid Y, Segre JA. The human skin microbiome. Nat Rev Microbiol. 2018 Mar;16(3):143-155. doi: 10.1038/nrmicro.2017.157. Epub 2018 Jan 15. PMID 29332945
- [Background] Aji, N., Kumala, S., Mumpuni, E., & Rahmat, D. (2022). Antibacterial Activity and Active Fraction of Zingiber officinale Roscoe, Zingiber montanum (J.Koenig) Link ex A., and Zingiber zerumbet (L.) Roscoe ex Sm. Against Propionibacterium acnes. Pharmacognosy Journal, 14(1), 103-111
- [Background] Kondapalli NB, Hemalatha R, Uppala S, Yathapu SR, Mohammed S, Venkata Surekha M, Rajendran A, Bharadwaj DK. Ocimum sanctum, Zingiber officinale, and Piper nigrum extracts and their effects on gut microbiota modulations (prebiotic potential), basal inflammatory markers and lipid levels: oral supplementation study in healthy rats. Pharm Biol. 2022 Dec;60(1):437-450. doi: 10.1080/13880209.2022.2033797. PMID 35188051
- [Background] Jaturapisanukul K, Udompataikul M, Kanokrungsee S, Rojhirunsakool S, Kamanamool N, Rachpirom M, Puttarak P. Efficacy and safety of a novel water-soluble herbal patch for acne vulgaris treatment: A randomized, assessor-blinds controlled, intra-individual split-face comparative study. Dermatol Ther. 2021 May;34(3):e14925. doi: 10.1111/dth.14925. Epub 2021 Mar 14. PMID 33651470
- [Background] Franco P, De Marco I. The Use of Poly(N-vinyl pyrrolidone) in the Delivery of Drugs: A Review. Polymers (Basel). 2020 May 13;12(5):1114. doi: 10.3390/polym12051114. PMID 32414187
- [Background] Elias AE, McBain AJ, O'Neill CA. The role of the skin microbiota in the modulation of cutaneous inflammation-Lessons from the gut. Exp Dermatol. 2021 Oct;30(10):1509-1516. doi: 10.1111/exd.14420. Epub 2021 Jul 11. PMID 34173265